CLINICAL TRIAL: NCT06456073
Title: An Open-Label, Single-Center, Investigator Initiated Phase 1B Trial of E-CEL UVEC Cell Therapy for the Treatment of Chronic Anal Fissure
Brief Title: E-CEL UVEC Treatment for Anal Fissures
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Angiocrine Bioscience (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-11026760
Record Dates: First submitted 2024-06-06; First posted 2024-06-13 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Chronic Anal Fissure
Keywords: Chronic Anal Fissure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention Arm (Experimental): Local percutaneous injection of E-CEL UVEC cells around the anal fissure
  Interventions: Biological: E-CEL UVEC cells (AB-207)

INTERVENTIONS:
Biological: E-CEL UVEC cells (AB-207) — Allogeneic (consented-maternal donor) E4ORF1+ (pro-survival gene transduced) human umbilical vein endothelial cells (percutaneous injection formulation)

SUMMARY:
This clinical trial is being conducted by investigators who are colorectal surgeons. Eligible study participants will receive the experimental treatment E-CEL UVEC cells by direct injection into the anal fissure. The study is being conducted to determine if E-CEL UVEC cell injections will be safe and would have any effects on healing of the anal fissure.

DETAILED DESCRIPTION:
This Phase 1b trial is conducted to evaluate the initial safety and efficacy of local (percutaneous) injections of E-CEL UVEC cells, genetically-engineered (pro-survival gene, E4ORF1+), human umbilical vein endothelial cells, as an experimental treatment of patients with chronic anal fissure (CAF) who have failed medical therapy (i.e., topical vasodilators ± botulinum injection). The study is a non-randomized, open-label, single arm study, meaning every study participant will receive some dose of the experimental study drug (no placebo). Consented, eligible participants will receive percutaneous injections of E-CEL UVEC cell product along the sides of the fissure; the treatments are spaced 3 to 4 weeks apart. Initial safety and efficacy parameters will be observed over a 6-month period, followed by a long-term follow-up consisting of annual questionnaire provided by electronic means.

This research study is being done because, in animal studies, E-CEL UVEC cells have been shown to aid in restoring or accelerating the normal healing in various tissues. This study will test if it is safe to use E-CEL UVEC cell therapy and if they it would aid in restoring or improve healing of CAF that was not responding to medical therapy. This study is being led by Dr. Kelly Garrett, Associate Professor of Surgery, and conducted by surgeons in the Colon and Rectal Surgery Division of Weill Cornell Medical College.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18 years and older
2. Anterior or posterior chronic anal fissure (CAF) - chronicity defined as presence of anal fissure ≥ 6 weeks
3. Inadequate response to medical treatment of anal fissure (1 month of failed vasodilator treatment plus declined or failed botulinum injection treatment)
4. Recent history of pain on defecation at a level 4 or higher on the numerical rating scale (NRS)
5. Vital signs upon screening:

   * Blood pressure: systolic ≥ 90 and < 140; and diastolic ≥ 60 and < 90.
   * Breathing: ≥ 12 and ≤ 20 breaths per minute.
   * Pulse: ≥ 60 and ≤ 100 beats per minute.
   * Temperature: ≥ 97.8°F and ≤ 99.1°F (36.5°C to 37.3°C)
   * O2 saturation: > 92%
6. Willing to take adequate contraceptive measures
7. Willing to sign an informed consent form and follow instructions for the trial including appearing for visits and filling out questionnaires

Exclusion Criteria:

1. Lateral anal fissure
2. Presence of peri-anal or rectovaginal fistula, rectal or anal stenosis, or peri-anal abscess or non-healing peri-anal post-surgical wounds that are not anal fissures (subjects with history of anorectal surgery with healed surgical wound is not excluded)
3. Active, untreated or medically unresponsive infection of the anal fissure or fistula (e.g., erythema and pus)
4. Active systemic infection (e.g., bacteremia, sepsis) - stable, controlled and treated HIV+ subjects (e.g., recent plasma HIV RNA <200 copies/mL) are not excluded
5. Presence of inflammatory bowel diseases (e.g., Crohn's, ulcerative colitis)
6. Taking systemic chemotherapy or local pelvic radiation treatments
7. Renal impairment defined by serum creatinine ≥ 1.5 x upper limit of normality (ULN)
8. Hepatic impairment defined by both of the following laboratory ranges:

   (a) total bilirubin ≥ 1.5 x ULN unless benign congenital hyperbilirubinemia; and (b) aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≥ 2.5 x ULN
9. Active alcohol or substance use that, in the opinion of the site investigator, will interfere with study follow-up.
10. Active malignant tumor (tumors must be in remission for ≥ 6 months without maintenance chemotherapy and/or radiation)
11. Ongoing or recent history (within 6 months) of abnormal, severe, progressive, or uncontrolled hepatic, hematological, gastrointestinal, endocrine, pulmonary, cardiac, neurological, psychiatric, or cerebral diseases
12. Congenital immunodeficiencies
13. History of major surgery or severe trauma within the previous 3 months
14. Subjects who are actively being considered as candidates for solid organ transplantation or who may have a high likelihood of needing a solid organ transplant (ex. Progressive heart failure)
15. Females who are pregnant or breastfeeding or planning to become pregnant or breastfeed during the study (180 days)
16. Subjects who have known hypersensitivity or documented allergy to DMSO
17. Subjects who do not wish to or cannot comply with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-09-12 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of severe injection site reactions | Up to 180 days
  Severe refers to Grade ≥ 3 as per CTCAE v5.0 terms and grading
Number of severe injection site reactions that are serious adverse events related to IP | Up to 180 days
Proportion of treated responders | Up to 180 days
  Treated responders is defined as ≥ 50% reduction in pain-on-defecation (using numerical rating scale (NRS)) and ≥ 50% reduction in fissure-wound area (based on clinical examination supplemented by photo-documentation) from baseline

SECONDARY OUTCOMES:
Changes in severity of pain on defecation (NRS) from (Day 0) baseline | Days 0, 14, 21, 28, 42, 56, 90 and 180
  Based on Numerical Rating Scale (NRS) measures at timepoints compared to baseline. Scale ranges from 0-10 with 0 representing no pain and severity of pain increasing chronologically.
Change in proportion of treated responders | Days 0, 14, 21, 28, 42, 56, 90 and 180
  Treated responders are defined as ≥ 50% reduction in pain-on defecation (using numerical rating scale (NRS)) and ≥ 50% reduction in fissure-wound-area (mm2) from baseline (Day 0)
Proportion of treated subjects who have complete cessation of fissure-related symptoms | Up to 180 days
Median percent change in fissure-wound from baseline (Day 0) | Days 0, 14, 21, 28, 42, 56, 90 and 180
  Median percent change in fissure wound size based on mm^2 using digital photo-image analysis
Mean percent change in fissure-wound from baseline (Day 0) | Days 0, 14, 21, 28, 42, 56, 90 and 180
  Mean percent change in fissure wound size based on mm^2 using digital photo-image analysis
Proportion of treated subjects who have ≥ 50% wound closure from baseline (Day 0) | Day 14
Proportion of treated subjects who have ≥ 50% wound closure from baseline (Day 0) | Day 21
Proportion of treated subjects who have ≥ 50% wound closure from baseline (Day 0) | Day 28
Proportion of treated subjects who have ≥ 50% wound closure from baseline (Day 0) | Day 42
Proportion of treated subjects who have ≥ 50% wound closure from baseline (Day 0) | Day 56
Proportion of treated subjects who have ≥ 50% wound closure from baseline (Day 0) | Day 90
Proportion of treated subjects who have ≥ 50% wound closure from baseline (Day 0) | Day 180
Time-to-response in days in treated responders | Up to 180 days
  Treated responders are defined as those with ≥50% reduction in pain on defecation (using numerical rating scale (NRS)) and ≥50% reduction in fissure-wound area from baseline (Day 0).
Time-to symptom improvement in days in treated subjects who achieved symptom improvement | Up to 180 days
  Symptom improvement is defined as a minimum 50% reduction in pain-on defecation (using numerical rating scale (NRS)) in treated subjects.
Time-to 50% wound closure in days in subjects who achieved at least 50% wound closure | Up to 180 days
Time-to complete wound closure in days in subjects who achieved complete wound closure | Up to 80
Cumulative number of severe adverse events, defined and graded by NCI CTCAE v5.0 | Up to 180 days
Percent of serious adverse events, including relatedness category | Up to 180 days
  Percent of SAE and relatedness categories of SAE as defined and graded by NCI CTCAE v5.0
Percent of treatment-emergent adverse events per system organ class (SOC) | Up to 180 days
Proportion of fissure relapse in treated subjects | Up to 180 days
  Fissure relapse is defined as worsening of pain and increase in size after healing.
Time-to-relapse in days in subjects who experienced relapse | Up to 180 days
  Days to relapse from time of healing.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Garrett, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No